CLINICAL TRIAL: NCT00043810
Title: Dose Finding Study of Gelonin Purging of Autologous Stem Cells for Transplantation of Patients With AML/MDS in First or Subsequent Remission
Brief Title: Study of Gelonin Purging of Autologous Stem Cells for Transplantation
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID02-060
Record Dates: First submitted 2002-08-14; First posted 2002-08-15 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Acute Myelogenous Leukemia; Myelodysplastic Syndrome
Keywords: AML; MDS; Gelonin; Purging; Transplant; Peripheral Stem Cell
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — GEL protein, Gelonium multiflorum; Busulfan; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gelonin Purging of ASCT (Experimental): Gelonin Purging of Autologous Stem Cells for Transplantation (ASCT) + Fludara/Busulfan
  Interventions: Procedure: Gelonin; Drug: Busulfan; Drug: Fludarabine

INTERVENTIONS:
Procedure: Gelonin — Gelonin-AntiCD33 purging, 3 purging concentrations (fixed dose of 5 x 10^6 CD34+ cells/kg to be infused) with 3 dose levels of 1 nanomolar, 5.0 nanomolar and 10.0 nanomolar.
  Other Names: HuM195-Gelonin conjugate
Drug: Busulfan — 130 mg/m2 in normal saline over three (3) hours IV every twenty-four (24) hours for four (4) consecutive days (days -6 to -3).
  Other Names: Busulfex; Myleran
Drug: Fludarabine — 40 mg/m2 in 100 ml of saline over one (1) hour on each of four (4) consecutive days (days - 6 to -3).
  Other Names: Fludara; Fludarabine Phosphate

SUMMARY:
Patients with Acute Myelogenous Leukemia or Myelodysplastic are able to achieve a complete remission but fail to achieve a prolonged disease-free survival. High dose chemotherapy and autologous bone marrow transplantation has been shown to be effective in this group of patients but hematopoietic recovery is slow, and infectious or bleeding complications are common. The delay in hematopoietic recover is accentuated by the use of purging techniques. This is a novel purging approach for autologous stem cell transplantation in patients with Acute Myelogenous Leukemia or Myelodysplastic syndrome to allow for rapid engraftment with a lower relapse rate therefore improving the therapeutic outcomes

DETAILED DESCRIPTION:
Treatment:

The HuM195-Gelonin conjugate has been designed to target leukemia cells and destroy them.

This treatment is divided into 3 parts.

Part I:

MOBILIZATION and STEM CELL COLLECTION:

This is the process that allows for collection of the autologous stem cells (the cells that will be used to do the transplant). All participants will receive the drug idarubicin by vein for 3 days together with cytarabine by vein for 3 days. This will be followed by injections of filgrastim (Neupogen) under the skin twice a day until the white count has recovered and the stem cells are collected. During the process, the number of stem cells in the blood will be measured. When the number of cells reach a certain level, participants will go through a collection procedure known as apheresis.

The apheresis procedure includes collecting blood through a large catheter placed under the collarbone or in the arm with the assistance of a device known as a cell separator. This device separates the stem cells from the rest of the blood and returns the rest of the blood to the participant. The procedure is usually done as an outpatient and takes between 4-5 hours to perform. Most patients collect enough cells for a transplant after 1 or 2 procedures. In this study, a maximum of 5 procedures are allowed.

Participants who are unable to have enough cells collected to take part in the study procedures, will be taken off study and offered alternative standard or investigational therapy. Participants will be able to leave the hospital with physician approval. They will then be monitored on a daily basis until the white blood cell count has recovered (usually 4-5 weeks). The stem cell collection can be done as either an inpatient or outpatient procedure depending on the participant's condition.

Part II:

PURGING PROCEDURE:

The stem cells that are collected through the apheresis procedure are treated in the laboratory with the Hum195/Gelonin conjugate. This procedure is known as purging and it is being studied to learn if the treatment of the stem cells with the HuM195/Gelonin conjugate can eliminate leukemia cells without damaging the normal stem cells. Since the best dose of HuM195/Gelonin conjugate for purging is not known, the cells of the participants in this study will receive 1 of 3 different doses of HuM195/Gelonin. The dose of HuM195/Gelonin that the cells will receive will be decided randomly according to the experience of the participants treated earlier in the study.

The first 3 participants in this study will receive cells that have not been treated with HuM195/Gelonin

After the cells have been treated, they are frozen for future use after the high dose busulfan treatment is given. As a safety measure, all participants will need to have a proportion of untreated stem cells as a back up. These can come from the original stem cell harvest or from a bone marrow harvest.

Part III:

HIGH DOSE FLUDARABINE/BUSULFAN WITH AUTOLOGOUS STEM CELL TRANSPLANT:

All participants who had enough cells treated with HuM195-Gelonin conjugate will then receive busulfan. Busulfan will be given by vein once a day for four days. It will be given together with fludarabine by vein once a day for 4 days. Three days after participants receive the last dose of busulfan, they will receive their previously stored stem cells through a blood transfusion. All participants will receive supportive care. This will include antibiotics, transfusions of blood products, extra nutrients, pain medication, and medications that will quicken the recovery of white blood cells. Participants will be on study for at least 12 months after the stem cell transplant coming for regular check ups.

All participants will have busulfan blood levels checked at specific times before, during and after busulfan infusion. On occasion more blood levels may be drawn. Levels are drawn through a small needle placed in the hands or arms of the patients and removed after the last busulfan blood draw. The busulfan dose administered MAY be modified according to the levels to prevent side effects. Two teaspoons of blood will be drawn for these measurements each time.

Participants will remain in the hospital for about 4-6 weeks and as an outpatient for 1 to 3 months. After participants leave the Medical Center Area, they will be seen in the transplant center every 3 to 6 months for 2 years.

This is an investigational study. The FDA has authorized the use of the HuM195-Gelonin conjugate in research only. Fludarabine has been previously approved for treatment of chronic lymphocytic leukemia by the FDA. The injectable solution of busulfan is a new preparation that has been approved by the FDA for allogeneic transplantation for chronic myelogenous leukemia (CML). The use of these drugs in this study is investigational. Up to 24 patients will be enrolled on this study. All will be enrolled at UTMDACC.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AML, RAEB-t, RAEB, or CMML who are in first remission and have poor prognosis cytogenetic abnormalities (i.e: deletions of chromosome 5, 7, 20; trisomy 8, t9,22,11q23 abnormalities or complex karyotypes).*
* Patients with AML, RAEB-t, RAEB, or CMML who are in second or subsequent remission.
* Remission is defined as ANC>1.5 x 109/Lt; Platelet count >100 x 109/Lt, and red cell transfusion independence.
* Male or female who have provided written informed consent.
* Tumor cells must be > 80 % CD-33 positive by flow cytometry.
* For women of childbearing potential (i.e., exclude post-menopausal women, women who have been surgically sterilized), adequate birth control methods must be used. Acceptable birth control methods are limited to oral contraceptives, implants, diaphragm, IUD or spermicide used with a condom)
* No chemotherapy for the two weeks prior to entering the study.
* No evidence of residual toxic effects from prior chemotherapy.
* Patients with proven bacterial infection are not eligible until resolution of the infection (patient afebrile, not on steroids). Patients with active fungal infections are eligible only if evidence of response to antifungal medications is documented and they do not have fever exceeding 38C.
* Must have at least 5 x 106 CD34+ peripheral blood stem cells collected.
* All patients who have had less than 7 x 106 CD34+ cells/kg collected, should have a bone marrow harvest to serve as back-up.
* A minimum of 1 x 106 CD34+ cells/kg of unpurged bone marrow or 2 x 106 CD34+ cells/kg of unpurged peripheral blood need to be stored as backup to be eligible for this protocol.
* Patients must have bilirubin less than 2.0, transaminases less than 4 x upper limit of normal.
* Pulmonary function tests >50% predicted for DLCO, FVC and FEV1
* No active uncontrolled infection
* No active CNS disease
* No uncontrolled arrythmias
* Zubrod Performance Status less than or equal to 2

Exclusion Criteria:

* Active CNS disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2002-07; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Optimal Dose Gelonin | 28 days post transplant
  Dose-finding success, defined as patient alive and engrafted at day 28 post transplant, represented as number of patient successes with 3 differing doses (5, 10, or 15 nanomolar (nm) gelonin-antiCD33 purged autologous stem cells after a high dose fludarabine/busulfan conditioning regimen).

CONTACTS AND LOCATIONS:
Overall Officials: Sergio A. Giralt, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org